CLINICAL TRIAL: NCT00816699
Title: Effects of Providing Preprint Preoperative Anesthetic Risk Information
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Effects of providing preprint preoperative anesthetic-risk information, Faculty of Medicine Siriraj hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Si325/2008
Record Dates: First submitted 2009-01-01; First posted 2009-01-05 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Preoperative Anxiety
Keywords: Anxiety; preprint anesthetic risk information
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Routine anesthetic risk information
  Interventions: Other: preprint preoperative anesthetic risk information
- 2 (Active Comparator): Preprint preoperative risk information
  Interventions: Other: preprint preoperative anesthetic risk information

INTERVENTIONS:
Other: preprint preoperative anesthetic risk information — preprint preoperative anesthetic risk information

SUMMARY:
Proportion of patients in study group(preprint preoperative anesthetic risk should have more anxiety, more knowledge, and more cancellation than controlled group

ELIGIBILITY:
Inclusion Criteria:

* Inpatients scheduled for surgery under general anesthesia with or without regional anesthesia
* Low to moderate risk surgery

Exclusion Criteria:

* Patient's refusal
* Patients scheduled for cardiovascular surgery and neurosurgery
* Patients with consciousness change following surgery
* Emergency case
* CNS or psychological diseases

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2008-12; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Spielberger State Trait Anxiety Inventory Scale | 5 days

SECONDARY OUTCOMES:
Knowledge, proportion of patients who cancel surgery, proportion who refuse regional anesthesia | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Suwannee Suraseranivongse, Principal Investigator — Department of Anesthesiology, Siriraj Hospital; Suwannee Suraseranivongse, MD, Principal Investigator — Department of Anesthesiology, Siriraj Hospital
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol Unversity, Bangkok, Thailand

REFERENCES:
- See also: Mahidol University — http://www.mahidol.ac.th